CLINICAL TRIAL: NCT03385889
Title: Effects of Cervical Spine Manual Therapy on Range of Motion, Joint Position Sense, and Balance in Participants With Cervicogenic Headache
Brief Title: Effects of Cervical Manual Therapy on Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenandoah University (Other)
Responsible Party: Principal Investigator, Aaron Hartstein, Assistant Professor of Physical Therapy, Shenandoah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShenandoahU(2017-2018)
Record Dates: First submitted 2017-12-20; First posted 2017-12-29 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Unilateral Headache; Musculoskeletal Neck Pain
Keywords: Cervicogenic Headache; Manual Therapy; Joint Position Sense; Balance
MeSH Terms: conditions — Headache; Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: Pre-test, Post-test, control group design 3 groups - mobilization, manipulation, control
Who Masked: Outcomes Assessor
Masking Description: Assessors of joint position sense, balance, and cervical spine range of motion via the Cervical Flexion Rotation Test will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cervical Spine Mobilization Group (Experimental): Subjects with cervicogenic headache who will be assigned to cervical spine mobilization group and receive intervention directed to C1/2 of ipsilateral side of unilateral dominant headache.
  Interventions: Procedure: Cervical Spine Mobilization
- Cervical Spine Manipulation Group (Experimental): Subjects with cervicogenic headache who will be assigned to cervical spine manipulation group and receive intervention directed to C1/2 of ipsilateral side of unilateral dominant headache.
  Interventions: Procedure: Cervical Spine Manipulation
- Control Group (No Intervention): No intervention. Subjects in this groups will wait for 5 minutes between pre- and post-testing of dependent variables.

INTERVENTIONS:
Procedure: Cervical Spine Mobilization — C1/2 graded mobilizations (Grade III/IV) provided to C1/2 segment on ipsilateral side of unilateral headache. Mobilizations will be completed for 3 sets of 30 seconds.
  Arms: Cervical Spine Mobilization Group
Procedure: Cervical Spine Manipulation — C1/2 manipulation (Grade V) provided to C1/2 segment on ipsilateral side of unilateral headache. The goal of the manipulation technique is to elicit an audible cavitation. If no cavitation is achieved upon the first attempt, a second and final attempt will be completed. No more than two attempts will be utilized per each subject in this allocated group.
  Arms: Cervical Spine Manipulation Group

SUMMARY:
The effects of cervical spine manual therapy, including mobilization and manipulation, on cervical spine range of motion, joint position sense, and balance is unknown among individuals with cervicogenic headache. Previous studies have indicated improved frequency of headache, decreased perceived disability, and demonstrated improved neuromuscular function following upper cervical manipulation. Other authors report improved cervical spine range of motion, joint position sense, and balance following cervical spine manual therapy for individuals with cervicogenic dizziness. Through an experimental design, this study aims to determine the effects of cervical spine manual therapy on variables such as cervical spine range motion, joint position sense, and balance among individuals with headache of a cervical spine origin.

DETAILED DESCRIPTION:
A convenience sample will be utilized to obtain subjects who suffer from cervicogenic headaches, as defined by the International Headache Classification. Subjects will be given an online medical screening questionnaire to differentiate and screen additional types of headache symptoms (migraine, cluster, tension-type, for example) and identify possible contraindications for manual therapy treatment techniques and exclude individuals if necessary. Subjects will be randomized into one of three groups (upper cervical mobilization, upper cervical manipulation, or control) and be tested with the Cervical Flexion Rotation Test, Joint Position Error testing, and sensorimotor balance testing via NeuroCom Balance Master. Subjects with cervicogenic headaches will receive their assigned intervention and dependent variables will be reassessed immediately, as well as 4-weeks after initial intervention. Individuals in either intervention group (mobilization or manipulation) will also complete a specific home-exercise program, which has been reported to improve upper cervical range of motion, to the C1/2 segment.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Signs and symptoms consistent with cervicogenic headache (including unilateral headache, headache that improves or resolves as cervical disorder or lesion improves or resolves, headache that is made worse with cervical movement or sustained painful neck positions, reduced cervical range of motion
* Headache frequency of at least once a week for 3 months

Exclusion Criteria:

* Bilateral headaches
* Non-musculoskeletal red flags
* Two or more positive neurologic signs indicative of nerve root compression
* Diagnosed with cervical spinal stenosis
* Bilateral upper extremity symptoms
* Symptoms indicative of central nervous system lesion
* History of whiplash injury within the previous 6 weeks
* Prior head or neck surgery
* Has received treatment for head or neck pain from any practitioner within the previous month
* Has received physical therapy or chiropractic treatment for head or neck pain within the previous 3 months
* Having a known vestibular or balance dysfunction (BPPV, unilateral vestibular loss, etc.)
* Other headaches that do not originate from the cervical spine, primarily migraine, vascular (cervical artery dysfunction), and tension-type headache.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Cervical Flexion Rotation Test (CFRT) | Post-Intervention, 4-weeks
  The Cervical Range of Motion (CROM) instrument will be placed on the subject. The subject will lie supine on the treatment table. The investigator will then passively flex the entire cervical spine and then rotate the head to both the left and right. The range of motion available in each direction, as measured by the CROM, will be recorded.

SECONDARY OUTCOMES:
Change in Joint Position Error | Post-Intervention, 4-weeks
  The subject will have a small laser pointer mounted onto a lightweight headband, which they will wear. The patient will be seated 90 cm from the wall. The starting point that is projected by the laser on the bullseye is marked. The patient will have their eyes closed and will perform an active neck movement. After this, the patient will return their head as accurately as possible to the starting position. This will include 6 trials, which will include cervical flexion, extension and rotation. The final laser position is measured against the starting position in centimeters. Errors will be measured following active return from cervical extension, flexion and rotation.
Change in Balance as measured by NeuroCom Balance Master | Post-Intervention, 4-weeks
  A pre-programmed option on the NeuroCom Balance Master will be utilized to assess the Modified Clinical test of Sensory Interaction on Balance (mCTSIB). Three different conditions will be utilized and each condition will last 30 secs. Three trials will be completed for each condition.First, the subject will be asked to maintain their balance while their eyes are closed. The amount of postural sway that they demonstrate will be recorded. Second, the subject will be asked to maintain their balance with their eyes open while the platform on the NeuroCom Balance Master force plate moves. The amount of postural sway demonstrated will be recorded. Third, the subject will be asked to rotate their head all the way to the left, then rotate their head all the way to the right. They will continue rotating between sides for the duration of the 30 second trial. The amount of postural sway that they demonstrate will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Abraham, PhD, PT, Study Director — Shenandoah University
Locations (1):
- Shenandoah University, Winchester, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Result] Dunning JR, Butts R, Mourad F, Young I, Fernandez-de-Las Penas C, Hagins M, Stanislawski T, Donley J, Buck D, Hooks TR, Cleland JA. Upper cervical and upper thoracic manipulation versus mobilization and exercise in patients with cervicogenic headache: a multi-center randomized clinical trial. BMC Musculoskelet Disord. 2016 Feb 6;17:64. doi: 10.1186/s12891-016-0912-3. PMID 26852024
- [Result] Reid SA, Callister R, Katekar MG, Rivett DA. Effects of cervical spine manual therapy on range of motion, head repositioning, and balance in participants with cervicogenic dizziness: a randomized controlled trial. Arch Phys Med Rehabil. 2014 Sep;95(9):1603-12. doi: 10.1016/j.apmr.2014.04.009. Epub 2014 May 2. PMID 24792139
- [Result] Kristjansson E, Treleaven J. Sensorimotor function and dizziness in neck pain: implications for assessment and management. J Orthop Sports Phys Ther. 2009 May;39(5):364-77. doi: 10.2519/jospt.2009.2834. PMID 19411769
- [Result] de Vries J, Ischebeck BK, Voogt LP, van der Geest JN, Janssen M, Frens MA, Kleinrensink GJ. Joint position sense error in people with neck pain: A systematic review. Man Ther. 2015 Dec;20(6):736-44. doi: 10.1016/j.math.2015.04.015. Epub 2015 May 2. PMID 25983238